CLINICAL TRIAL: NCT00894205
Title: Neuropsychological and Physiological Effects of Low-Impact Exercise for Older Adults
Brief Title: Neuropsychological Effects of Strengthening Exercise for Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Union College, New York (Other)
Responsible Party: Principal Investigator, Cay Anderson-Hanley, Associate Professor, Union College, New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2078
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Cognitive Ability, General
Keywords: neuropsychological function; cognitive function; exercise; older adult
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- strengthening exercise (Experimental): A low intensity strengthening exercise program based on the Tufts University "Strong Bones" program. Utilizes small free weights and chair exercises.
  Interventions: Behavioral: strengthening exercise program

INTERVENTIONS:
Behavioral: strengthening exercise program — A low intensity strengthening exercise program based on the Tufts University "Strong Bones" program. Utilizes small free weights and chair exercises. Participants attend community based class 2-3x/wk for 4 wks.
  Other Names: Strong Bones

SUMMARY:
This study aims to examine the benefits to thinking processes of a low intensity, strengthening exercise program for older adults.

DETAILED DESCRIPTION:
The neuropsychological benefits, especially executive function impacts, of four weeks of a low intensity, strengthening exercise program will be examined for community residing older adults.

ELIGIBILITY:
Inclusion Criteria:

* independent living
* older adult
* interested in strengthening exercise program

Exclusion Criteria:

* must meet Strong Bone's screening criteria or have physician's approval

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Function | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cay Anderson-Hanley, PhD, Principal Investigator — Union College
Locations (1):
- Strong Bones community class locations, Schenectady, New York, United States